CLINICAL TRIAL: NCT05090878
Title: AtheroGEnic LipoprotEinS in Ischemic Stroke: The AGELESS Study
Brief Title: Atherogenic Lipoproteins in Ischemic Stroke
Acronym: AGELESS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01167; ko21Demarchis2
Record Dates: First submitted 2021-10-06; First posted 2021-10-25 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Ischemic Stroke
Keywords: Apolipoprotein B (apoB); Lipoprotein(a) (Lp(a)); Low-density Lipoprotein Cholesterol (LDL-C); Very Low-density Lipoprotein (VLDL); Intraplaque Hemorrhage (IPH); Atherogenic lipoproteins; Dyslipidemia
MeSH Terms: conditions — Ischemic Stroke; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological material (blood) in this project is not identified by participant name but by a unique participant number. Biological material is appropriately stored in a restricted area only accessible to authorized personnel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1. Patients with and without carotid IPH: Among patients with carotid artery atherosclerosis (stenosis 30-99%), patients with and without IPH, as assessed by MR-Plaque Imaging, are compared in terms of apoB, Lp(a) levels and other cardiovascular risk factors.
- 2. Patients with and without first-ever ischemic stroke at baseline: Among patients with carotid artery atherosclerosis (stenosis 30-99%), the risk of first-ever ischemic stroke in relation to apoB, Lp(a) levels, and presence of IPH is assessed, after adjusting for the cardiovascular factors.
- 3. Patients with and without recurrent ischemic stroke: Among patients with carotid artery atherosclerosis (stenosis 30-99%) with an ipsilateral ischemic stroke at baseline, the risk of recurrent ipsilateral ischemic stroke in relation to apoB, Lp(a) levels, and presence of IPH is assessed, after adjusting for the cardiovascular factors.

SUMMARY:
Apolipoprotein B (apoB) levels (which encompass all atherogenic lipoproteins, including LDL), Lp(a) levels, and carotid IPH are associated with both first-ever and recurrent ischemic stroke.

This cohort research project is to analyze:

1. Among patients with carotid artery atherosclerosis (stenosis 30-99%), to compare patients with and without IPH, as assessed by magnetic resonance (MR)-Plaque Imaging, in terms of apoB, Lp(a) levels and other cardiovascular risk factors. (IPH is a strong morphological sign of plaque vulnerability / instability and a strong marker of consecutive atheroembolic events).
2. Among patients with carotid artery atherosclerosis (stenosis 30-99%), to assess the risk of first-ever ischemic stroke in relation to apoB, Lp(a) levels, and presence of IPH, after adjusting for the cardiovascular factors (understanding this association can inform primary prevention).
3. Among patients with carotid artery atherosclerosis (stenosis 30-99%) with an ipsilateral ischemic stroke at baseline, to assess the risk of recurrent ipsilateral ischemic stroke in relation to apoB, Lp(a) levels, and presence of IPH, after adjusting for the cardiovascular factors. There will be a sensitivity analysis to assess if the association between Lp(a) and recurrent stroke is stronger in patients <60 years of age. (understanding this association can inform secondary prevention).

For the first and second aim, there will be a cross-sectional, case-control analysis. For the third aim, i.e. assessing recurrent ischemic stroke, there is prospective follow-up of at least 3 months up to 45 months.

ELIGIBILITY:
Inclusion Criteria:

* Atherosclerotic carotid stenosis, North American Symptomatic Trial Collaborators (NASCET) method 30-99%
* Ability to undergo a neck MR for carotid plaque imaging
* Ability to undergo a follow-up of at least 1-year
* For the prospective, longitudinal part: Hemispheric ischemic stroke or retinal ischemia ipsilateral to the carotid stenosis, with symptom onset within 24 hours (these patients will be followed-up for recurrent ischemic stroke)

Exclusion Criteria:

* Carotid stenosis due to causes other than atherosclerosis (e.g. carotid dissection or post-actinic)
* Contraindication to MRI
* Lack of informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke will be recruited in the Stroke Unit of the University Hospital Basel (primary center) and Zurich (partner center). Patients without ischemic stroke will be recruited in the outpatient neurovascular clinic at the University Hospital Basel (primary center) and Zurich (partner center), where around 250 patients with known carotid stenosis are regularly followed-up - clinically and with ultrasound.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Presence of carotid IPH on MR-Plaque imaging (3-Tesla MR scans with an 8-channel carotid coil) | one time assessment at baseline (scan time is 5 minutes)
  Presence of carotid IPH on MR-Plaque imaging at baseline. Baseline means either acquired during the hospitalization for the index stroke or during the enrolling visit at the outpatient consultation of the neurovascular clinic of the University Hospital Basel (primary center) and Zurich (partner center).
Presence of an ischemic, hemispheric, ipsilateral stroke on baseline brain MR-Diffusion Weighted Imaging (DWI) | one time assessment at baseline
  Presence of an ischemic, hemispheric, ipsilateral stroke, i.e. on the same side of the carotid stenosis, on baseline brain MR-DWI.
Presence of a recurrent ischemic, hemispheric, ipsilateral stroke in the 3-month follow-up brain MR-DWI | 3 months after baseline
  Presence of a recurrent ischemic, hemispheric, ipsilateral stroke in the 3-month follow-up brain. The 3-month follow-up brain MR-DWI is conceived to detect covert strokes, i.e. clinically asymptomatic strokes, as recurrences tend to occur short after the first stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Gian Marco De Marchis, PD Dr. med., Principal Investigator — Department of Neurology/Stroke Center; University Hospital Basel
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Department of Neurology/Stroke Center, Basel
  - University Hospital Zürich, Zurich